CLINICAL TRIAL: NCT07352579
Title: From Screening to Support: A Multi-Method Analysis of HRSN Integration in Cancer Care
Status: Recruiting | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: iRISID-2025-1005; JT 46229 (Other: JeffTrial Number)
Record Dates: First submitted 2026-01-09; First posted 2026-01-20 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Cancer
Keywords: Health-Related Social Needs; HRSNs; transportation access; food insecurity; housing instability; utility needs; Survey; Interview
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer Patients Screened for Health-Related Social Needs (HRSNs): This group includes adult cancer patients receiving care at Sidney Kimmel Comprehensive Cancer Center (SKCCC) who previously completed a Health-Related Social Needs (HRSNs) screening in the electronic health record. This will be achieved by providing patients with a one-time survey. The surveys will be distributed via MyChart messages and emails. Additionally, 20 patients who complete the survey will be asked to complete a short interview to further understand why cancer patients identified as high-risk for HRSNs decline connections to care and intervention-ultimately to gain an understanding into the factors that they take into account when determining whether they want to be connected to a resource or service connection related to HRSNs.
  Interventions: Other: Survey; Other: Interview

INTERVENTIONS:
Other: Survey — Participants complete a one-time electronic survey to assess factors influencing the decision to decline assistance for identified Health-Related Social Needs (HRSNs). The survey includes questions related to transportation access, food insecurity, housing instability, and utility needs. Survey completion takes approximately 10 minutes.
Other: Interview — Interviews will be semi-structured and will be offered to 20 participants who have completed the survey and meet eligibility criteria. Interviews will be conducted via a Zoom. Zoom will create a transcription of the interview which will be saved in a secure encrypted space, no video will be saved.

SUMMARY:
This observational study aims to identify the factors that influence whether cancer patients accept or decline supportive care services after screening positive for health-related social needs (HRSNs) at the Sidney Kimmel Comprehensive Cancer Center.

The study focuses on adult oncology patients who previously reported at least one HRSN-such as transportation, food, housing, or utility needs-but declined assistance when it was offered.

The main questions it aims to answer are:

* What factors shape cancer patients' intentions to use supportive care services for HRSNs?
* Why do patients who screen positive for HRSNs choose not to accept help offered by the healthcare system?

Participants will:

* Complete a one-time electronic survey delivered via MyChart or email.
* Optionally participate in a semi-structured Zoom interview (for a subset of 20-30 survey respondents) to explore decision-making in greater depth.

DETAILED DESCRIPTION:
This is a cross-sectional observational study. There will be 500 participants for MyChart survey and 20 participants for semi-structured interviews. Surveys will be distributed via MyChart and email and will take about 10 minutes to complete. The main purpose of this study is to understand why SKCCC participants are not seeking support for their corresponding HRSNs from the healthcare system. The hypothesis is that a range of factors are contributing to SKCCC patients' decline of resources to address risks identified in HRSN screening potentially inclusive of mistrust of healthcare systems, perception that there are no resources to help, feelings others can use the resources more than themselves, as well as protective factors like past resiliency and resourcefulness. An examination of the initial HRSN screening data for cancer patients within this health system revealed that, in 2024, 5,727 (74.7%; n=7662) patients who were in active cancer treatment completed the HRSN screening questionnaire in four domains: transportation access, food insecurity, housing instability, and utility needs. Of these, 716 patients (12.5%) reported having a need in at least one HRSN domain. However, only 343 patients (47.9%, n = 716) wanted help from the healthcare system to address their HRSN(s). This highlights that the majority (52.1%, n = 716) of cancer patients in active treatment who have been screened for HRSN have unmet needs that could be addressed but are not being flagged as such in our healthcare system. This preliminary data sheds light on the concrete and resource needs of cancer patients, but there is not a good understanding of why participants are not seeking support for their corresponding HRSNs from the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must meet all of the following inclusion criteria in order to be eligible to participate in the study:

  * Provide informed consent via check box for survey
  * Provide verbal consent via Zoom for interview
  * Must be able to read and understand English
  * Willing to comply with all study procedures and be available for the duration of the study
  * Patients with existing HRSN data in their EHR that answere4d yes to risk in at least one domain and no to wanting help/follow up

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in this study:

  * If they do not consent
  * Non-patients with existing HRSN data in their EHR
  * Individuals unable to complete the survey due to language barriers or other cognitive limitations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult cancer patients who received care at SKCCC who were engaged in HRSN screening
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Factors influencing cancer patients' intent to use oncology supportive care for HRSNs | approximately 4 months
  Measured via Surveys (self-reported) using a structured questionnaires with binary (Yes/No) responses and Likert Style questions (Quality of Life and FACT-ES).

SECONDARY OUTCOMES:
Factors associated with declining HSRN-related supportive care services | approximately 4 months
  Interviews will be semi-structured and will be offered to 20 participants who have completed the survey and meet eligibility criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Munjireen Sifat, PhD, MPH, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States